CLINICAL TRIAL: NCT04867018
Title: Defining the Pathophysiology of Heterotopic Ossification: A Prospective Study
Status: Withdrawn | Type: Observational
Why Stopped: study was never fully reopened with the intuitional review board
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jon Schoenecker, Associate Professor Of Orthopaedics, Pathology, Pharmacology, and Pediatrics, Vanderbilt University Medical Center
Other Study IDs: 333333
Record Dates: First submitted 2021-03-19; First posted 2021-04-30 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Heterotopic Ossification
MeSH Terms: conditions — Ossification, Heterotopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Orthopaedic Trauma, Pediatrics and Joint Patients: Patients will have an additional 9ml of blood drawn during their normal course of care for this study up to 4 times. Intraoperatively, we will request a tissue sample of the debrided injured muscle from the area where the surgeon is operating. There will be no additional tissue sample taken during the surgery, but what is removed in the normal course of the operation will be used for analysis in our study.
- Healthy Volunteer: Blood will be taken from healthy, nonpregnant adults who weigh at least 110 pounds. All volunteers will have a single blood draw of 100ml at the time of consent.

SUMMARY:
Our overarching aim is to define the pathophysiology, epidemiology, and natural history of HO by following patients from date of injury until full wound healing has occurred and the window for HO has passed.

Specific aims

Aim 1: To classify the acute and chronic physiologic profiles of fracture patients and how they relate to the development of HO. Here the investigators will look at the systemic derangements to patients' coagulation, fibrinolytic, and inflammatory profiles.

Aim 2: Identify the true incidence and time course of HO development after traumatic fracture. To accomplish this the investigators will look at patients who have sustained hip fracture, midshaft/distal femur fracture, humerus fracture, proximal radius fracture, and elbow dislocation/fractures and track follow-up images up to one year after injury looking for HO.

Aim 3: Define the histologic characteristics of HO development. To accomplish this aim the investigators will perform a histologic analysis on a sample of injured muscle surrounding the fracture area.

Aim 4: To determine what comorbid, iatrogenic, or environmental influences are associated with the formation of HO. To achieve this aim the investigators will evaluate data including injury type, surgery type, operative duration, surgical approach, contamination (open vs closed injury), complications (malunion, nonunion, infection, hardware failure, removal of hardware), hardware type, comorbidities (smoking, cardiac history, diabetes), and medications.

DETAILED DESCRIPTION:
The aforementioned general inclusion/exclusion criteria will be used to determine patient eligibility. All eligible patients will be identified using a patient list from StarPanel provided by the managing team. The study will proceed until all eligible patients are enrolled (our goal for this study is to recruit at least 1000 patients). If the patient agrees to participate in the study they will be asked to sign an informed consent document by the research team.

Arm 1

On Admission:

Demographics and Comorbidities The following patient data will be recorded: age, gender, height, weight, date of admission, date of discharge, diagnosis, injury time, injury type, laterality, surgical approach, implants used, duration of surgery, time to union, contamination (open vs closed injury), comorbidities (smoking, cardiac history, diabetes, etc.), current medications.

Labs Patients will have an additional 9ml of blood drawn during their normal course of care for this study up to 4 times. The draws will happen while they are an inpatient in the hospital. The timing of the draw will surround the timing of their operation. They will have blood drawn within 24 hours before surgery, immediately after surgery, 24 hours after surgery, and 72 hours after surgery. Labs values, including CBC with dif, CMP, D-Dimer, CRP, PT/INR, PTT, fibrinogen, lactate, PAI-1, plasminogen activation assay, chromogenics, plasmin-anti-plasmin complex, and phosphate will be collected for this study. Patient often have a blood draw before and after surgery, one for typing and another as part of routine labs. The investigators will use the remnants of those blood draws which will be stored in the Vanderbilt Lab core and retrieved for further analysis by key research personnel. The remaining plasma will come from another remnant blood or an extra draw.

Tissue Samples Intraoperatively, investigators will request a tissue sample of the debrided injured muscle from the area where the surgeon is operating. There will be no additional tissue sample taken during the surgery, but what is removed in the normal course of the operation will be used for analysis in our study. The amount of tissue that will be analyzed for this study will vary based on how much of the injured muscle the operating physician decides to take in their normal course of operation. If the tissue sample is not readily accessible, such as in the case of an intramedullary nail fixation, the investigators will forgo the sample.

Follow-up

Radiographic imaging and notes from follow-up appointments will be examined for complications, such as: malunion, nonunion, infection, hardware failure, removal of hardware, presence of amorphous tissue calcification, symptomatic HO, or asymptomatic HO. Time to the development of calcific complications, will also be recorded. To document post-surgical complications the investigators will use imaging, photographs, progress notes, clinic notes, ICD-9 codes, CPT codes and operative reports.

The time frame for follow up visits will be based on the preference of the participant's physician. Any complications resulting from the injury will be documented. Complications will be documented if they occur within 2 years of injury. No study activities will take place during this time frame other than recording complications.

Clinical Practice Guidelines

All patients will be treated according to established clinical practice guidelines at Vanderbilt Children's Hospital or Vanderbilt Medical Center, decreasing the chance that differences in the patients' results and outcomes result from variability of the treating physician.

Arm 2 Volunteers Blood Draw Blood will be taken from healthy, nonpregnant adults who weigh at least 110 pounds. All volunteers will have a single blood draw of 100ml at the time of consent. No more than 2.5% of the volunteer's blood volume will be taken at any point (100ml maximum for a 110lb person in one sitting).

ELIGIBILITY:
Arm 1- Injured Patients

Inclusion Criteria:

* Any patient treated in our hospital system from initial IRB approval until we reach our enrollment quota that are diagnosed with HO, hip fracture, midshaft/distal femur fracture, humerus fracture, proximal radius fracture, and elbow dislocation/fracture. This includes patients in all age groups and of all genders.
* Patients with a diagnosis of HO, hip fracture, midshaft/distal femur fracture, humerus fracture, proximal radius fracture, or elbow fracture must be receiving operative treatment for their injury.
* Patients with concurrent trauma will be grouped into a sub-analysis.

Exclusion Criteria:

* Patients with pathologic fractures.
* Non-operative patients other than elbow dislocation patients
* Pregnant Women
* Patients who do not intend to follow-up at Vanderbilt

Arm 2- Healthy Volunteers

Inclusion Criteria:

* Volunteers (male or female) between ages of 18-70
* Weight greater than 110lbs

Exclusion Criteria:

* Chronic medical conditions such as diabetes, hypertension, high cholesterol, rheumatologic disorders, infections, etc.
* History of recent trauma or burn injury
* Recent inpatient admission within the last year
* Pregnant females or people on hormone replacement therapy
* People on any anticoagulant medication or NSAIDS

Max Age: 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Injured patients will be recruited from the orthopedic trauma, pediatrics and joints service from clinics.
  Healthy volunteers will be solicited from flyers around the VUMC medical center and through ResearchMatch.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Change of coagulation from baseline during hospitalization as measured by platelet count | Change of platelet count from baseline and during hospitalization (approximately 1-28 days)
  The normal platelet count range is 150,000-450,000/uL. Typically a decrease in platelet count is associated with activation of coagulation, and increases represent a rebound reparative period. This is not always the case, so we will record both increases and decreases in platelet count, specifically.
Change of coagulation from baseline during hospitalization as measured by thrombin-antithrombin (TAT) complexes | Change of thrombin-antithrombin (TAT) from baseline and during hospitalization (approximately 1-28 days)
  The normal range for thrombin-antithrombin (TAT) complexes is 1-4 ug/L. An increase in thrombin-antithrombin (TAT) complexes will indicate activation of coagulation.
Change of fibrinolysis from baseline during hospitalization as measured by plasmin-antiplasmin complex (PAP) | Change of plasmin-antiplasmin complex (PAP) from baseline and during hospitalization (approximately 1-28 days)
  The normal range for Plasmin-antiplasmin complex (PAP) is 120-700ug/L. An increase in plasmin-antiplasmin complex (PAP) will indicate activation of fibrinolysis.
Change of fibrinolysis from baseline during hospitalization as measured by D-dimer | Change of D-dimer from baseline and during hospitalization (approximately 1-28 days)
  The normal range for D-dimer is <0.5mg/L. An increase in D-dimer will indicate activation of fibrinolysis.
Change of inflammation from baseline during hospitalization as measured by C-reactive protein (CRP) | Change of C-reactive protein (CRP) from baseline and during hospitalization (approximately 1-28 days)
  The normal range for C-reactive protein (CRP) is <10mg/L. An increase in C-reactive protein (CRP) will indicate activation of inflammation.
Change of inflammation from baseline during hospitalization as measured by IL-6 | Change of IL-6 from baseline and during hospitalization (approximately 1-28 days)
  The normal range for IL-6 is 0-5pg/mL or <15pg/mL. An increase in IL-6 will indicate activation of inflammation.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt Children's Orthopaedics, Nashville, Tennessee, United States